CLINICAL TRIAL: NCT01419938
Title: Does CBT Improve the Effect of Light Therapy in Delayed Sleep Phase Syndrome Compared to Only Light Therapy - Short and Long Term Follow up
Brief Title: Does Cognitive Behaviour Therapy (CBT) Improve the Effect of Light Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Uppsala County Council, Sweden (Other Government)
Responsible Party: Principal Investigator, Katarina Danielsson, M.D. Ph.D student., Uppsala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011/167
Record Dates: First submitted 2011-07-26; First posted 2011-08-18 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Delayed Sleep Phase Syndrome
Keywords: Light therapy; circadian rhythm; CBT
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm | interventions — Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Light therapy for two weeks (Active Comparator)
  Interventions: Device: Light therapy
- Light therapy and CBT (Active Comparator): Two weeks of light therapy and after that 4 weeks of Cognitive behaviour therapy (CBT)
  Interventions: Device: Light therapy and Cognitive behaviour therapy

INTERVENTIONS:
Device: Light therapy and Cognitive behaviour therapy — Light therapy every morning during 30 minutes for two weeks. CBT for 90 to 120 minutes weekly during four weeks.
  Arms: Light therapy and CBT
Device: Light therapy — Light therapy every morning during 30-45 minutes for two weeks.
  Arms: Light therapy for two weeks

SUMMARY:
Delayed sleep phase syndrome (DSPS) is the most common of the circadian rhythm sleep disorders (CRSD). A person with DSPS have sufficient sleep quality, but their circadian clock is delayed compared to the normal 24-h period. They fall asleep around 03.00-04.00 at night and sleeps until 02.00-03.00 in the afternoon. This syndrome is most frequent among young people between 16-25 years, which conveys that school attendance and education are affected, and also often results in severe social consequences. DSPS is sometimes associated with depression and personality disorders and may aggravate psychiatric symptoms.

This syndrome is highly underdiagnosed and there are no detailed guidelines how to treat it. The treatment usually consists of light therapy, chronotherapy or melatonin. There is a lack of guidelines how often, with which wavelength, and how long the treatment of DSPS patients shall go on. Previous studies shows that light therapy often is effective. The effect gets even better if melatonin is administered concurrently. However, the frequency of relapse is high.

Thus, DSPS is a prevalent syndrome in young adults with severe consequences on normal daytime functioning. There are almost no treatment options available in health care settings. There is a clear need for further studies on this topic. The main purpose of the present study is to evaluate the clinical effects of short and long-term treatment by using light therapy and cognitive behaviour therapy (CBT). CBT is recommended at mild to moderate depression and anxiety. It also has some evidence in treating insomnia. Patients with DSPS often have al of these symptoms and therefore the investigators would like to investigate if CBT can enhance the effect of light therapy.

Firstly, the investigators want to evaluate the short-term effects of light therapy with and without CBT. Secondly, the investigators want to evaluate if the patients who get CBT maintain a "normal" sleep rhythm and prevent relapse of DSPS compared to just light therapy for two weeks.

The investigators also want to evaluate how this patient-group differs when it comes to behavioral factors compared to a matched reference group.

DETAILED DESCRIPTION:
DSPS patients delayed sleep and wake times are accompanied by insomnia and excessive sleepiness that results in functional impairments. The sleeping-problems and the impairment in important areas of functioning and quality of life sometimes lead to psychiatric problems such as, depressive symptoms, irritability, problems with their memory and concentration. It has not yet been fully established how long the treatment should go on, how long each light treatment should be, and the exact intensity of light. Although long-term studies on DSPS patients are sparse, it is known from clinical experience that these patients often fall back into their old circadian schedule after the treatment.

This study is a prospective randomised study. In the short-term study patients will be randomised to two groups. Group I light therapy (LT) for two weeks Group II LT for two weeks + CBT for four weeks. Group I and II will be followed up with questionnaires concerning depression/anxiety, sleepiness during the day, sleep-diary and insomnia-problems.

The aim is to evaluate if CBT enhance LT-treatment at home. The two groups will be followed with sleep-diary monthly and questionnaires.

Method. Questionnaires. All patients will fill in some questionnaires before the treatment starts, during treatment and at follow-up.

I) Horne-Ostberg Morning-Eveningness Questionnaire (MEQ) to measure their diurnality.

II) Insomnia Severity Scale (ISI), a scale that measures the severity of insomnia III) Epworth Sleepiness Scale (ESS), a scale that measures habitual daytime sleepiness.

IV) Hospital anxiety- depression scale (HADS) V) Penn state Worry Questionnaire (PSWQ) VI)Symptom-focused Rumination Scale (SRS) VII) Brief COPE(BC) The same questionaires will be given to a matched reference group, but without sleeping problems.

Light therapy: It is today considered that the most effective light intensity is 10 000 lux at approximately one foot from the person and during 30-45 minutes. This treatment will be applied at home. The exact time schedule for the light treatment will be decided individually depending on the patient's sleep diary. Each day the time for light therapy will be brought back one hour earlier and thereby getting out of bed.

CBT will be given for 90-120 minutes by a psychologist once per week for four weeks at our Sleep Department. The therapy will be given in groups of 4-6 persons.

DLMO. DLMO will only be taken before the study starts to evaluate the shift in circadian rhythm. DLMO is the time when endogenous melatonin reaches a threshold of 3 ng/L or 4 ng/L in saliva. To measure melatonin in saliva is the most commonly used way to determine DLMO since it is both easy and safe for the patient and it gives a value that follows the melatonin blood-value, only it is three times lower. The saliva test will be taken hourly for about five hours, during a window when we suspect DLMO to appear. It is important that the saliva collection must be done under dim light conditions (less then 10 lux).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of delayed sleep phase syndrome.

Exclusion Criteria:

* Eye diseases
* Active psychiatric disorder.
* Ongoing somatic disorder.

Ages: 16 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2011-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in sleep-diary at 6 months. | Change from baseline in sleep-diary at 6 months.
  That the patients will go to bed before 01:00 and wake up not later than 09:00 a.m. or earlier.

SECONDARY OUTCOMES:
Changes from baseline in sleep-diary at 6 weeks. | Changes from baseline in sleep diary at 6 weeks.
  That the patients will go to bed before 01:00 and wake up not later than 09:00 a.m. or earlier.
Change from baseline in Hospital anxiety-depression scale at 2 weeks | Change from baseline in Hospital anxiety-depression scale at 2 weeks
  By comparing the results of the questionnaires before study start, during and after study completion. Knowledge about this patient group will provide clinical routines to treat patients with DSPS. The results will also be compared with a matched reference-group.
Change from baseline in Hospital anxiety-depression scale at 6 weeks | Change from baseline in Hospital anxiety-depression scale at 6 weeks
  By comparing the results of the questionnaires before study start, during and after study completion. Knowledge about this patient group will provide clinical routines to treat patients with DSPS. The results will also be compared with a matched reference-group.
Change from baseline in Hospital anxiety-depression scale at 6 months | Change from baseline in Hospital anxiety-depression scale at 6 months
  By comparing the results of the questionnaires before study start, during and after study completion. Knowledge about this patient group will provide clinical routines to treat patients with DSPS. The results will also be compared with a matched reference-group.
Change from baseline in Insomnia Severity Scale at 2 weeks | Change from baseline in Insomnia Severity Scale at 2 weeks
  By comparing the results of the questionnaires before study start, during and after study completion. Knowledge about this patient group will provide clinical routines to treat patients with DSPS. The results will also be compared with a matched reference-group.
Change from baseline in Insomnia Severity Scale at 6 weeks | Change from baseline in Insomnia Severity Scale at 6 weeks
  By comparing the results of the questionnaires before study start, during and after study completion. Knowledge about this patient group will provide clinical routines to treat patients with DSPS. The results will also be compared with a matched reference-group.
Change from baseline in Insomnia Severity Scale at 6 months | Change from baseline in Insomnia Severity Scale at 6 months
  By comparing the results of the questionnaires before study start, during and after study completion. Knowledge about this patient group will provide clinical routines to treat patients with DSPS. The results will also be compared with a matched reference-group.
Change from baseline in Epworth Sleepiness Scale at 2 weeks | Change from baseline in Epworth Sleepiness Scale at 2 weeks
  By comparing the results of the questionnaires before study start, during and after study completion. Knowledge about this patient group will provide clinical routines to treat patients with DSPS. The results will also be compared with a matched reference-group.
Change from baseline in Epworth Sleepiness Scale at 6 weeks | Change from baseline in Epworth Sleepiness Scale at 6 weeks
  By comparing the results of the questionnaires before study start, during and after study completion, knowledge about this patient group will provide clinical routines to treat patients with DSPS. The results will also be compared with a matched reference-group.
Change from baseline in Epworth Sleepiness Scale at 6 months | Change from baseline in Epworth Sleepiness Scale at 6 months
  By comparing the results of the questionnaires before study start, during and after study completion. Knowledge about this patient group will provide clinical routines to treat patients with DSPS. The results will also be compared with a matched reference-group.
Change from baseline in Penn State Worry Questionnaire at 6 months | Change from baseline in Penn State Worry Questionnaire at 6 months
  By comparing the results of the questionnaire before study start and after study completion. Knowledge about this patient group will provide clinical routines to treat patients with DSPS. The results will also be compared with a matched reference-group.
Change from baseline in Symptom-focused Rumination Scale at 6 months | Change from baseline in Symptom-focused Rumination Scale at 6 months
  By comparing the results of the questionnaire before study start and after study completion. Knowledge about this patient group will provide clinical routines to treat patients with DSPS. The results will also be compared with a matched reference-group.
Change from baseline in Brief COPE at 6 months | Change from baseline in Brief COPE at 6 months
  By comparing the results of the questionnaire before study start and after study completion. Knowledge about this patient group's coping strategies will provide clinical routines to treat patients with DSPS. The results will also be compared with a matched reference-group.
Change from baseline in sleep-diary at 2 weeks | Change from baseline in sleep-diary at 2 weeks
  That the patients will go to bed before 01:00 and wake up not later than 09:00 a.m. or earlier
Number of participants that will keep their new sleep-timings. | 6 months
  We want to measure how many participants that can keep their new sleep-timings after the first treatment (6 weeks). We believe that CBT or light-therapy intermittently can help these patients to avoid relapses
Change from baseline in Horne-Ostberg Morning-Eveningness Questionnaire at 6 months | Change from baseline in Horne-Ostberg Morning-Eveningness Questionnaire at 6 months
  By comparing the results of the questionnaire before study start and after study completion. Knowledge about this patient group will provide clinical routines to treat patients with DSPS. The results will also be compared with a matched reference-group.

OTHER OUTCOMES:
Does DLMO correlate with sleep diary | baseline
  A part of a second study. About the importance of DLMO. Since DLMO has been measured in this patient group at baseline
Is DLMO important for setting the time to start light therapy | From baseline to 2 weeks
  Is a sleep diary enough or is DLMO important to decide the time to start Light therapy in the morning.
Is scores in MEQ important to decide when to start light therapy in the morning. | from baseline to 2 weeks of Light therapy
  Is scores in MEQ important to decide when to start light therapy in the morning. and are scores in MEQ correlated with DLMO and sleep diary

CONTACTS AND LOCATIONS:
Overall Officials: Katarina ML Danielsson, M.D., Principal Investigator — Sleep department, Uppsala University Hospital, Sweden; Agneta Markstroem, Ass. Prof., Principal Investigator — Sleep department, Uppsala University Hospital, Sweden; Jan-Erik Broman, Ass. Prof., Principal Investigator — Sleep department, Uppsala University Hospital, Sweden; Markus Jansson-Fröjmark, Ass. Prof., Principal Investigator — Department of Psychology, Stockholm University, Sweden
Locations (1):
- Sleep department, Uppsala, Sweden

REFERENCES:
- [Background] Benloucif S, Burgess HJ, Klerman EB, Lewy AJ, Middleton B, Murphy PJ, Parry BL, Revell VL. Measuring melatonin in humans. J Clin Sleep Med. 2008 Feb 15;4(1):66-9. PMID 18350967
- [Background] Gooley JJ. Treatment of circadian rhythm sleep disorders with light. Ann Acad Med Singap. 2008 Aug;37(8):669-76. PMID 18797560
- [Background] Bjorvatn B, Pallesen S. A practical approach to circadian rhythm sleep disorders. Sleep Med Rev. 2009 Feb;13(1):47-60. doi: 10.1016/j.smrv.2008.04.009. Epub 2008 Oct 8. PMID 18845459
- [Background] Dagan Y, Yovel I, Hallis D, Eisenstein M, Raichik I. Evaluating the role of melatonin in the long-term treatment of delayed sleep phase syndrome (DSPS). Chronobiol Int. 1998 Mar;15(2):181-90. doi: 10.3109/07420529808998682. PMID 9562922